CLINICAL TRIAL: NCT00702351
Title: A Phase II, Uncontrolled Pilot Trial to Evaluate That a Single Dose of 100 μg or 150 μg Org 36286 (Corifollitropin Alfa) is Able to Induce Multiple Follicular Growth During the First Week of Controlled Ovarian Stimulation for IVF or ICSI Using a Long Protocol of GnRH Agonist (Study 38833)
Brief Title: A Trial of Single Dose Corifollitropin Alfa's Ability to Induce Multiple Follicular Growth During the First Week of Controlled Ovarian Stimulation for IVF or ICSI (38833)(P05788)
Acronym: Realize
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P05788; EudraCT #: 2004-004968-68;; 38833
Record Dates: First submitted 2008-06-18; First posted 2008-06-20 (Estimated); Last update posted 2022-02-02 (Actual); Status verified 2022-02

CONDITIONS: In Vitro Fertilization
Keywords: Infertility; Pharmacological effects of drugs; Drug therapy; Hormones; GnRH agonist; RecFSH; Corifollitropin alfa; Open-label
MeSH Terms: conditions — Infertility | interventions — follicle stimulating hormone, human, with HCG C-terminal peptide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): 150 µg Org 36286 (corifollitropin alfa)
  Interventions: Drug: Org 36286 (corifollitropin alfa)
- Arm 2 (Experimental): 100 µg Org 36286 (corifollitropin alfa)
  Interventions: Drug: Org 36286 (corifollitropin alfa)

INTERVENTIONS:
Drug: Org 36286 (corifollitropin alfa) — A single dose of Org 36286 will be administered after down-regulation has been confirmed (E2 below 50 ng/L and P below 1.48 μg/L). The first group comprising subjects weighing >= 50 kg will receive a dose of 150 μg Org 36286 (150 μg dose group). The second group comprising subjects weighing <= 60 kg will receive a dose of 100 μg Org 36286 (100 μg dose group).
  Other Names: corifollitropin alfa

SUMMARY:
To evaluate the induction of multiple follicular growth after single dose administration of 100 μg or 150 μg Org 36286 in a long protocol of GnRH agonist.

DETAILED DESCRIPTION:
In this trial, all subjects were (pre)treated daily with subcutaneous triptorelin, a GnRH agonist which is known to provide profound suppression of endogenous LH and FSH. It was evaluated whether these down-regulated subjects show an appropriate ovarian response to 100 μg or 150 μg Org 36286 during the first week of stimulation. To evaluate this, follicular growth was measured by USS, and serum inhibin-B and E2 levels were assessed.

ELIGIBILITY:
Inclusion Criteria:

* Females of couples with an indication for controlled ovarian stimulation (COS) and IVF or ICSI that have had at least one previous COS cycle with proven normal ovarian response;
* >=18 and <= 39 years of age at the time of signing informed consent;
* a. First group: Body weight >= 50 kg and BMI >= 18 and <= 29 kg/m^2; b. Second group: Body weight <= 60 kg and BMI <= 29 kg/m^2;
* Normal menstrual cycle length: 24-35 days;
* Ejaculatory sperm (use of donated and/or cryopreserved sperm is allowed);
* Normal routine diagnostic hysteroscopy and endometrial biopsy;
* Willing and able to sign informed consent.

Exclusion Criteria:

* History of or any current (treated) endocrine abnormality;
* History of ovarian hyper-response1 or history of ovarian hyperstimulation

syndrome (OHSS);

* History of or current polycystic ovary syndrome (PCOS);
* A basal antral follicle count > 20 (size < 11 mm, both ovaries combined) on USS during the early follicular phase (menstrual cycle day 2-5);
* Less than 2 ovaries or any other ovarian abnormality;
* Presence of unilateral or bilateral hydrosalpinx (visible on USS);
* Presence of unilateral or bilateral endometriomas (>10 mm; visible on USS);
* More than three unsuccessful COS cycles since the last established ongoing

pregnancy (if applicable);

* History of non- or low ovarian response to FSH/hMG treatment;
* FSH or LH > 12 IU/L as measured by the local laboratory (sample taken during the early follicular phase: menstrual cycle day 2-5);
* Any clinically relevant abnormal laboratory value based on a sample taken during the screening phase;
* Contraindications for the use of gonadotropins (e.g. tumors, pregnancy/lactation, undiagnosed vaginal bleeding, hypersensitivity, ovarian cysts) or GnRH analogues (e.g. hypersensitivity, pregnancy/lactation);
* Recent history of or current epilepsy, diabetes or cardiovascular, gastro-intestinal, hepatic, renal or pulmonary disease;
* History or presence of alcohol or drug abuse within 12 months prior to signing informed consent;
* Previous use of Org 36286;
* Use of hormonal preparations within 1 month prior to screening;
* Administration of investigational drugs within three months prior to signing

informed consent.

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2005-12-09 (Actual); Primary Completion 2007-03-26 (Actual); Study Completion 2007-07-11 (Actual)

PRIMARY OUTCOMES:
serum inhibin-B levels; follicle number and follicle size distribution | One cycle

SECONDARY OUTCOMES:
Amount of recFSH needed from Stimulation Day 8 onwards to the Day of hCG; Endocrinological parameters (FSH, LH, E2, P); Number and quality of oocytes retrieved | One cycle
Number of fertilized oocytes; Fertilization rate; Number and quality of embryos; Implantation rate; Miscarriage rate; Clinical outcome | One cycle

REFERENCES:
- [Result] Fatemi HM, Oberye J, Popovic-Todorovic B, Witjes H, Mannaerts B, Devroey P. Corifollitropin alfa in a long GnRH agonist protocol: proof of concept trial. Fertil Steril. 2010 Oct;94(5):1922-4. doi: 10.1016/j.fertnstert.2009.12.070. Epub 2010 Feb 10. PMID 20149360